CLINICAL TRIAL: NCT02190123
Title: REalWorld Insights on the INitiation and Treatment Duration of ticagrEloR & Other Oral Antiplatelets in Patients With Acute Coronary Syndrome in Belgium/Luxembourg (REWINDER)
Brief Title: REalWorld Insights on the INitiation and Treatment Duration of ticagrEloR & Other Oral Antiplatelets (OAP) in Patients With Acute Coronary Syndrome (ACS) in Be/Lux.
Acronym: REWINDER
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-CBE-XXX-2014/1
Record Dates: First submitted 2014-07-11; First posted 2014-07-15 (Estimated); Last update posted 2016-01-08 (Estimated); Status verified 2016-01

CONDITIONS: Treatment of Acute Coronary Syndrome (ACS).
Keywords: Acute Coronary Syndrome (ACS); Oral antiplatelets (ticagrelor, prasugrel, clopidogrel) (OAP); Treatment persistence.
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — OAP protocol

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ACS patients treated with OAP: Patients with ACS who have been initiated and treated with ticagrelor and other oral antiplatelets
  Interventions: Drug: ACS patients treated with OAP

INTERVENTIONS:
Drug: ACS patients treated with OAP — Patients with ACS who have been initiated and treated with ticagrelor and other oral antiplatelets.

SUMMARY:
REWINDER is a multinational, multicentre, non-interventional, retrospective study of patients treated with an oral antiplatelet (ticagrelor, prasugrel or clopidogrel) while in hospital after an acute coronary syndrome (ACS) event, to be conducted in Belgium and Luxembourg.

Primary objective is to evaluate the actual treatment persistence with oral antiplatelets (OAP) after an ACS in the clinical practice in Belgium and Luxembourg.

The main secondary objectives are to describe the most frequent reasons for OAP treatment switch, discontinuation or reinitiation; to identify the decisionmakers in the OAP treatment changes and to characterize the patient profile in terms of demographics, diagnosis, management strategies, comorbidities and concomitant medications to identify any association between patient profile and treatment duration.

DETAILED DESCRIPTION:
Treatment of acute coronary syndrome (ACS) with oral antiplatelets (OAPs) is recommended for up to 12 months unless discontinuation is clinically indicated. Early discontinuation could result in an increased risk of cardiovascular death or myocardial infarction due to the patient's underlying disease.

There are no robust data allowing to evaluate the treatment persistence with OAPs after ACS in the current practice in Belgium and Luxembourg at this time. It is currently unclear as to why patients discontinue, switch or reinitiate treatment and upon whose advice. A non-interventional study is needed to obtain reliable data on treatment persistence and reasons for discontinuation, switch or reinitiation of treatment.

REWINDER is a multinational, multicentre, non-interventional, retrospective study of patients treated with an oral antiplatelet (ticagrelor, prasugrel or clopidogrel) while in hospital after an ACS event, to be conducted in Belgium and Luxembourg. Primary objective is to evaluate the actual treatment persistence with OAPs after an ACS in the clinical practice in Belgium and Luxembourg. The main secondary objectives are to describe the most frequent reasons for OAP treatment switch, discontinuation or reinitiation; to identify the decisionmakers in the OAP treatment changes and to characterize the patient profile in terms of demographics, diagnosis, management strategies, comorbidities and concomitant medications to identify any association between patient profile and treatment duration.

The target sample size of the study is 500 patients.

ELIGIBILITY:
Inclusion Criteria:

The patient population that will be observed in the NIS must fulfil all of the following criteria:

1. Female or male aged ≥18 years
2. A patient information letter has been sent by the Investigator to the patient
3. Patient discharged alive from this hospital to home following ACS (diagnosed with STEMI, NSTEMI or UA)
4. ACS is either UA or myocardial infarction of Type 1 (spontaneous myocardial infarction related to ischemia due to a primary coronary event such as plaque erosion and/or rupture, fissuring, or dissection)
5. ACS after 1st July 2012 and before 1st June 2013
6. Patient on ticagrelor, prasugrel or clopidogrel treatment at discharge following an ACS

Exclusion Criteria:

Patients will not be eligible to participate if any of the following exclusion criteria are present:

1. Patient who participated in any interventional clinical study during the observation period.
2. Patient with ACS precipitated by or as complication of surgery, trauma, gastrointestinal bleeding or after Percutaneous Coronary Intervention (PCI)
3. Patient with ACS occurring during a stay in the hospital

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female patients from Belgium and Luxembourg, aged 18 years or more , discharged alive from hospital to home following an acute coronary syndrome (ACS) and who were treated with an oral antiplatelet (OAP) (ticagrelor, prasugrel or clopidogrel) after an acute coronary syndrome (ACS) event (Unstable Angina (UA), ST-elevation myocardial infarction (STEMI) or non-STEMI(NSTEMI)).
Sampling Method: Non-Probability Sample
Enrollment: 430 (Actual)
Dates: Start 2014-09; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
The actual treatment persistence with OAP after an ACS in the clinical practice of Belgium and Luxembourg will be assessed by analysing the patient's 1-year follow data after discharge of an ACS event from hospital. Analysis will be descriptive. | up to 1 year
  Patients discharged after an ACS event and fulfilling the entry criteria will be included in each centre. The retrospective observation period will be 1 year, starting on the date of discharge to home. Data on OAD treatment situation during the observation period will be collected. Number and proportion of patients having stopped treatment after 1, 3, 6, 9 & 12 month will be assessed and described.

SECONDARY OUTCOMES:
The reasons for OAP treatment switch, discontinuation or re-initiation will be assessed by analysing the patient's 1-year follow data after discharge of an ACS event from hospital. Analysis will be descriptive. | up to 1 year
  Patients discharged after an ACS event and fulfilling the entry criteria will be included in each centre. The retrospective observation period will be 1 year, starting on the date of discharge to home. Data on OAD treatment situation during the observation period will be collected. The reasons for switch, discontinuation & re-initiation (side-effects, drug-drug interactions, cost of treatment, patient's complaint, high bleeding risk & other) will be assessed and described.

OTHER OUTCOMES:
The decisionmakers in the oral antiplatelet (OAP) treatment changes will be identified by analysing the patient's 1-year follow data after discharge of an ACS event from hospital. Analysis will be descriptive. | up to 1 year
  Patients discharged after an ACS event and fulfilling the entry criteria will be included in each centre. The retrospective observation period will be 1 year, starting on the date of discharge to home. Data on OAD treatment situation during the observation period will be collected. The decisionmakers will be identified and described (cardiologist interventional, cardiologist non interventional, surgeon, other specialist, dentist, GP, patient and/or family, other).
The patient profile will be characterized by analysing the patient's 1-year follow data after discharge of an ACS event from hospital. Analysis will be descriptive. | up to 1 year
  Patients discharged after an ACS event and fulfilling the entry criteria will be included in each centre. The retrospective observation period will be 1 year, starting on the date of discharge to home. Data on OAD treatment situation during the observation period will be collected. Patient profile will be described in terms of demographics, diagnosis, management strategies, comorbidities and concomitant medications to identify any association between patient profile and treatment duration.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Claeys, Prof Dr, Principal Investigator — Universitair Ziekenhuis Antwerpen (UZA)
Locations (15):
- Belgium (15):
  - Research Site, Aalst
  - Research Site, Baudour
  - Research Site, Bonheiden
  - Research Site, Brasschaat
  - Research Site, Bruges
  - Research Site, Brussels
  - Research Site, Charleroi
  - Research Site, Edegem
  - Research Site, Ghent
  - Research Site, Leuven
  - Research Site, Liège
  - Research Site, Mechelen
  - Research Site, Montegnée
  - Research Site, Ronse
  - Research Site, Uccle

REFERENCES:
- See also: Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=3037&filename=Synopsis.pdf